CLINICAL TRIAL: NCT07020728
Title: Speech Intelligibility and Listening Effort
Brief Title: Clarity in Motion Phase-1 Perceptual Study of Speech Intelligibility
Acronym: CIM PhI PercX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Speech Technology and Applied Research Corp. (Industry)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CIM Phase 1; 1R43DC020690-01A1 (NIH)
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Subjects in each arm heard different treatments (interventions) of the same set of target words (spondees). Subjects in all arms heard the same spondees (but with different treatments), and subjects in all arms heard stimuli with all treatments (but different spondees).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Group 1A (Experimental): Subjects in this Group listened and responded to a unique set of stimulus/treatment pairs.
  Interventions: Behavioral: Solo: Unmasked Speech Stimuli; Behavioral: Raw: Fully masked speech--no motion stimuli; Behavioral: StatScrub: Extracted Speech--no motion stimuli; Behavioral: SlideSpch: Scrubbed Speech emitted from linearly moving speaker stimuli; Behavioral: SlideNoise: Speech Scrubbed from linearly moving and stationary noise stimuli; Behavioral: SlideMic: Stationary sources scrubbed from a linearly moving mic stimuli
- Group 1B (Experimental): Subjects in this Group listened and responded to a unique set of stimulus/treatment pairs.
  Interventions: Behavioral: Solo: Unmasked Speech Stimuli; Behavioral: Raw: Fully masked speech--no motion stimuli; Behavioral: StatScrub: Extracted Speech--no motion stimuli; Behavioral: SlideSpch: Scrubbed Speech emitted from linearly moving speaker stimuli; Behavioral: SlideNoise: Speech Scrubbed from linearly moving and stationary noise stimuli; Behavioral: SlideMic: Stationary sources scrubbed from a linearly moving mic stimuli
- Group 2A (Experimental): Subjects in this Group listened and responded to a unique set of stimulus/treatment pairs.
  Interventions: Behavioral: Solo: Unmasked Speech Stimuli; Behavioral: Raw: Fully masked speech--no motion stimuli; Behavioral: StatScrub: Extracted Speech--no motion stimuli; Behavioral: SlideSpch: Scrubbed Speech emitted from linearly moving speaker stimuli; Behavioral: SlideNoise: Speech Scrubbed from linearly moving and stationary noise stimuli; Behavioral: SlideMic: Stationary sources scrubbed from a linearly moving mic stimuli
- Group 2B (Experimental): Subjects in this Group listened and responded to a unique set of stimulus/treatment pairs.
  Interventions: Behavioral: Solo: Unmasked Speech Stimuli; Behavioral: Raw: Fully masked speech--no motion stimuli; Behavioral: StatScrub: Extracted Speech--no motion stimuli; Behavioral: SlideSpch: Scrubbed Speech emitted from linearly moving speaker stimuli; Behavioral: SlideNoise: Speech Scrubbed from linearly moving and stationary noise stimuli; Behavioral: SlideMic: Stationary sources scrubbed from a linearly moving mic stimuli
- Group 3A (Experimental): Subjects in this Group listened and responded to a unique set of stimulus/treatment pairs.
  Interventions: Behavioral: Solo: Unmasked Speech Stimuli; Behavioral: Raw: Fully masked speech--no motion stimuli; Behavioral: StatScrub: Extracted Speech--no motion stimuli; Behavioral: SlideSpch: Scrubbed Speech emitted from linearly moving speaker stimuli; Behavioral: SlideNoise: Speech Scrubbed from linearly moving and stationary noise stimuli; Behavioral: SlideMic: Stationary sources scrubbed from a linearly moving mic stimuli
- Group 3B (Experimental): Subjects in this Group listened and responded to a unique set of stimulus/treatment pairs.
  Interventions: Behavioral: Solo: Unmasked Speech Stimuli; Behavioral: Raw: Fully masked speech--no motion stimuli; Behavioral: StatScrub: Extracted Speech--no motion stimuli; Behavioral: SlideSpch: Scrubbed Speech emitted from linearly moving speaker stimuli; Behavioral: SlideNoise: Speech Scrubbed from linearly moving and stationary noise stimuli; Behavioral: SlideMic: Stationary sources scrubbed from a linearly moving mic stimuli
- Group 4A (Experimental): Subjects in this Group listened and responded to a unique set of stimulus/treatment pairs.
  Interventions: Behavioral: Solo: Unmasked Speech Stimuli; Behavioral: Raw: Fully masked speech--no motion stimuli; Behavioral: StatScrub: Extracted Speech--no motion stimuli; Behavioral: SlideSpch: Scrubbed Speech emitted from linearly moving speaker stimuli; Behavioral: SlideNoise: Speech Scrubbed from linearly moving and stationary noise stimuli; Behavioral: SlideMic: Stationary sources scrubbed from a linearly moving mic stimuli
- Group 4B (Experimental): Subjects in this Group listened and responded to a unique set of stimulus/treatment pairs.
  Interventions: Behavioral: Solo: Unmasked Speech Stimuli; Behavioral: Raw: Fully masked speech--no motion stimuli; Behavioral: StatScrub: Extracted Speech--no motion stimuli; Behavioral: SlideSpch: Scrubbed Speech emitted from linearly moving speaker stimuli; Behavioral: SlideNoise: Speech Scrubbed from linearly moving and stationary noise stimuli; Behavioral: SlideMic: Stationary sources scrubbed from a linearly moving mic stimuli
- Group 5A (Experimental): Subjects in this Group listened and responded to a unique set of stimulus/treatment pairs.
  Interventions: Behavioral: Solo: Unmasked Speech Stimuli; Behavioral: Raw: Fully masked speech--no motion stimuli; Behavioral: StatScrub: Extracted Speech--no motion stimuli; Behavioral: SlideSpch: Scrubbed Speech emitted from linearly moving speaker stimuli; Behavioral: SlideNoise: Speech Scrubbed from linearly moving and stationary noise stimuli; Behavioral: SlideMic: Stationary sources scrubbed from a linearly moving mic stimuli
- Group 5B (Experimental): Subjects in this Group listened and responded to a unique set of stimulus/treatment pairs.
  Interventions: Behavioral: Solo: Unmasked Speech Stimuli; Behavioral: Raw: Fully masked speech--no motion stimuli; Behavioral: StatScrub: Extracted Speech--no motion stimuli; Behavioral: SlideSpch: Scrubbed Speech emitted from linearly moving speaker stimuli; Behavioral: SlideNoise: Speech Scrubbed from linearly moving and stationary noise stimuli; Behavioral: SlideMic: Stationary sources scrubbed from a linearly moving mic stimuli
- Group 6A (Experimental): Subjects in this Group listened and responded to a unique set of stimulus/treatment pairs.
  Interventions: Behavioral: Solo: Unmasked Speech Stimuli; Behavioral: Raw: Fully masked speech--no motion stimuli; Behavioral: StatScrub: Extracted Speech--no motion stimuli; Behavioral: SlideSpch: Scrubbed Speech emitted from linearly moving speaker stimuli; Behavioral: SlideNoise: Speech Scrubbed from linearly moving and stationary noise stimuli; Behavioral: SlideMic: Stationary sources scrubbed from a linearly moving mic stimuli
- Group 6B (Experimental): Subjects in this Group listened and responded to a unique set of stimulus/treatment pairs.
  Interventions: Behavioral: Solo: Unmasked Speech Stimuli; Behavioral: Raw: Fully masked speech--no motion stimuli; Behavioral: StatScrub: Extracted Speech--no motion stimuli; Behavioral: SlideSpch: Scrubbed Speech emitted from linearly moving speaker stimuli; Behavioral: SlideNoise: Speech Scrubbed from linearly moving and stationary noise stimuli; Behavioral: SlideMic: Stationary sources scrubbed from a linearly moving mic stimuli

INTERVENTIONS:
Behavioral: Solo: Unmasked Speech Stimuli — Speech stimuli recorded using non-moving speakers and mics. No masking sources present. No BSS applied to multi-channel recordings. Very high output QoS values.
  Other Names: Treat1
Behavioral: Raw: Fully masked speech--no motion stimuli — Speech stimuli recorded using non-moving speakers and mics. All masking sources present. No speech separation or extraction methods applied to multi-channel recordings. Very low output QoS values.
  Other Names: Treat2
Behavioral: StatScrub: Extracted Speech--no motion stimuli — Speech stimuli recorded using non-moving speakers and mics. All masking sources present. Joint ACES scrubbing of both noise sources applied to multi-channel recordings. Very high output QoS values.
  Other Names: Treat3
Behavioral: SlideSpch: Scrubbed Speech emitted from linearly moving speaker stimuli — Speech stimuli recorded using linearly moving speech source and stationary masking sources and mics. All masking sources present. Joint ACES scrubbing of both noise sources applied to multi-channel recordings. Moderately high output QoS values.
  Other Names: Treat4
Behavioral: SlideNoise: Speech Scrubbed from linearly moving and stationary noise stimuli — Mixed speech and noise sources recorded using a stationary speech source, a stationary noise source, and a linearly moving noise source. A valid source hypothesis of the speech source is used to extract the speech source. High output QoS values.
  Other Names: Treat5
Behavioral: SlideMic: Stationary sources scrubbed from a linearly moving mic stimuli — Mixed speech and noise sources recorded using all stationary sources, and a linearly moving microphone (mic 1). Joint ACES scrubbing of both noise sources is used to reduce the response of Mic 1 to a residue of speech. Low output QoS values.
  Other Names: Treat6

SUMMARY:
Participants received a bilateral pure-tone hearing screen administered by the research team. All potential participants who failed the hearing screen were provided with information about its meaning and referral for further audiological testing.

Participants who passed the hearing screen and other inclusion criteria were divided into 6 groups, each of which were presented with 144 stimuli equally distributed among processing conditions. Listeners choose a comfortable listening level using supplied headphones and were able to control the rate of presentation. Following a short practice session, listeners were be asked to transcribe each target sentence. The intelligibility of each stimulus was estimated by determining the mean percentage of content words correctly transcribed. After transcription, listeners were asked for two qualitative judgments: (1) the "clarity" of the stimulus, and (2) the "listening effort" involved. The quality of each stimulus was estimated by the median quality judgment, and the effort likewise. Listening sessions were located in a quiet room and presentation was controlled by the Superlab presentation software program.

The Stimuli consisted of audio recordings of target spondaic words embedded in a carrier sentence produced by a male and a female native speaker of American English recorded under quiet conditions. Each stimulus presented to the listeners for identification was either unmasked pristine speech or speech that had been processed in one of five ways with different mixtures of noise and sensor movement. The latter are identified as QoS Levels 1-5.

Collectively, the estimates of word intelligibility, clarity, and listening effort under the different conditions shed light on the effectiveness with which the tested algorithm preserves listener intelligibility with acceptable effort and quality.

DETAILED DESCRIPTION:
Participants received a bilateral pure-tone hearing screen administered by a clinically trained member of the research team. The threshold criteria was 20 dB SPL at 250 and 500 Hz, and 25 dB SPL at 1000, 2000, 4000, and 8000 Hz. All potential participants who failed the hearing screen were provided with information about its meaning and referred for further audiological testing.

Participants who passed the hearing screen and other inclusion criteria were divided into 6 groups, each of which was presented with 144 stimuli equally distributed among processing conditions (Pristine Non-Moving Speech plus QoS Levels 1-5). Listeners self-selected a comfortable listening level using supplied headphones and were able to control the rate of presentation. Following a short practice session, listeners were asked to transcribe the target sentences, and the intelligibility of each stimulus was estimated by determining the mean percentage of content words correctly transcribed. After transcription, listeners were also asked for two qualitative judgments using a visual analog scale: (1) the "clarity" of the stimulus, and (2) the "listening effort" involved. These measures are sensitive to situations where listeners manage to extract the uttered words from the signal, but with increasing difficulty. The quality of each stimulus was estimated by the median quality judgment, and the effort likewise. Listening sessions took place in a quiet room and presentation was controlled by the Superlab presentation software program.

The Stimuli consisted of audio recordings of target spondaic words embedded in a carrier sentence produced by a male and a female native speaker of American English recorded under quiet conditions. Each stimulus presented to the listeners for identification was either unmasked pristine speech or speech that had have been processed in one of five ways with different mixtures of noise and sensor movement. The latter are identified as QoS Levels 1-5. Each type of processing was expected to have a different effect on the underlying probability that the listener would be able to correctly identify the spoken word, the effort required to do so, and the quality of the presented recording. Data on familiarity ratings for the target spondaic words and relative intelligibility of the two speakers under different conditions of noise masking has been previously reported.

Collectively, the estimates of word intelligibility, clarity, and listening effort under the different conditions is expected to shed light on the effectiveness with which the tested algorithm preserves listener intelligibility with acceptable effort and quality.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will include adult native speakers of American English with auditory thresholds within age-normal limits, defined as passing a pure tone screening test of 20 dB SPL at 250 and 500 Hz, and 25 dB SPL at 1000, 2000, 4000, and 8000 Hz. Exclusion criteria will include self-report of hearing difficulties and failure to pass hearing screen.

No special populations requiring special protections will be utilized in this study. Potential participants who fail the hearing screen will be provided with results and appropriate clinical referral as per the IRB protocol.

Exclusion Criteria:

* Exclusion criteria will include self-report of hearing difficulties and failure to pass hearing screen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Target Word Transcription Accuracy | The subject transcribed the target word immediately after hearing the carrier phrase.
  For each audio stimulus of a target word in a carrier phrase, the subject transcribed the target word they heard (by typing that word in a field in the display. Their transcription was later graded as correct or incorrect by a researcher.
Listening Effort | Immediately after hearing the carrier phrase.
  Subject-reported effort required to identify word in carrier phrase, reported by moving a slider on a 0% to 100% scale.
Naturalness of speech | Immediately after hearing the carrier phrase.
  Subject-reported perceived naturalness of target word in carrier phrase, reported by moving a slider on a 0% to 100% scale.

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Goldhor, PhD, Principal Investigator — Speech Technology & Applied Research Corp.
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States